CLINICAL TRIAL: NCT05606406
Title: Hypoxia and Heart Rate Variability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Trishul Siddharthan, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220794
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Hypoxia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Control Group (Active Comparator): Individuals without lung disease will receive oxygen for a period of four hours
  Interventions: Other: Nocturnal Oxygen
- Nocturnal hypoxemia group (Active Comparator): Individuals with lung disease will receive oxygen for a period of four hours
  Interventions: Other: Nocturnal Oxygen

INTERVENTIONS:
Other: Nocturnal Oxygen — Nocturnal oxygen will be increased hourly for a period of four hours up to 4 liters per minute (LPM). If the oxygen saturation (SpO2) falls below 70% the oxygen rate will be increased until patients achieve the threshold of 70% and then will proceed with titrations of 1 liter per minute LPM per hour.

SUMMARY:
The purpose of this study is to evaluate how variations in oxygen demands may change heart electrical activity in individuals with and without oxygen dependence.

ELIGIBILITY:
Healthy Participants

Inclusion Criteria:

• Ability to provide consent

Exclusion Criteria:

* BMI > 40 kg/m2
* Prevalent myocardial infarction, coronary revascularization, heart failure, and stroke
* Unstable medical conditions that may preclude enrollment in the protocol such as: uncontrolled angina and/or congestive heart failure, uncontrolled blood pressure or resistant hypertension, cancer, and active psychiatric disease (e.g., major depression)

Nocturnal Hypoxemia

Inclusion Criteria:

* Ability to provide consent
* Chronic respiratory condition resting Sat < 95% off oxygen

Exclusion Criteria:

* BMI > 40 kg/m2
* Prevalent myocardial infarction, coronary revascularization, heart failure, and stroke
* Unstable medical conditions that may preclude enrollment in the protocol such as: uncontrolled angina and/or congestive heart failure, uncontrolled blood pressure or resistant hypertension, severe chronic obstructive pulmonary disease, cancer, and active psychiatric disease (e.g., major depression)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
QT Variability Index | Up to 10 hours
  Measured from electrocardiogram (ECG)

SECONDARY OUTCOMES:
Normalized variance of the heart rate (HRVN) | Up to 10 hours
  Measured from ECG
QT-RR interval | Up to 10 hours
  Measured from ECG

CONTACTS AND LOCATIONS:
Overall Officials: Trishul Siddharthan, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No